CLINICAL TRIAL: NCT00652366
Title: A Randomized, Open-label, Dose-escalation to Rash Study to Assess the Effect of Tarceva in Combination With Gemcitabine on Overall Survival in Patients With Metastatic Pancreatic Cancer.
Brief Title: A Dose-Escalation to Rash Study of Tarceva (Erlotinib) Plus Gemcitabine in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO21128; 2007-003751-37
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Results first posted 2015-02-11 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-01

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Erlotinib Hydrochloride; Gemcitabine

ARMS (2):
- Gemcitabine, Erlotinib Standard Dose (Active Comparator): Participants received erlotinib, 100 milligrams (mg), orally (PO), once daily until disease progression or unacceptable toxicity. Participants also received gemcitabine, 1000 mg per (/) square meter (m^2), intravenously (IV), on Days 1, 8, and 15 of consecutive 4 week cycles until disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib, standard dose; Drug: Gemcitabine
- Gemcitabine, Erlotinib Escalating Dose (Experimental): Participants received erlotinib, beginning at 150 mg/day, PO, once daily, and increasing in increments of 50 mg every 2 weeks up to a maximum of 250 mg/day, until development of a grade 2 rash, or occurrence of other, non-rash, dose-limiting toxicity; treatment was continued until disease progression, unacceptable toxicity, death or withdrawal. Participants also received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of consecutive 4 week cycles until disease progression or unacceptable toxicity.
  Interventions: Drug: Erlotinib, escalating dose; Drug: Gemcitabine

INTERVENTIONS:
Drug: Erlotinib, escalating dose — 100mg, PO, once daily, escalating to a maximum of 250mg, PO, once daily
  Other Names: Tarceva
  Arms: Gemcitabine, Erlotinib Escalating Dose
Drug: Erlotinib, standard dose — 100mg, PO, once daily
  Other Names: Tarceva
  Arms: Gemcitabine, Erlotinib Standard Dose
Drug: Gemcitabine — 1000 mg/m2, IV, on days 1,8 and 15 of each 4 week cycle

SUMMARY:
This study will compare the efficacy and safety of escalating versus standard doses to rash of Tarceva, in combination with gemcitabine, in patients with metastatic pancreatic cancer. During a 4 week run-in period, all patients will receive Tarceva 100mg/day po plus gemcitabine 1000mg/m2 iv on days 1, 8,15 and 22. After 4 weeks, patients who have not developed rash, or only develop grade 1 rash, will be randomized to one of 2 groups. Group 1 will receive a starting dose of Tarceva 150mg po daily, increased in steps of 50mg every 2 weeks up to a maximum of 250mg/day po, until development of grade 2 rash or other dose-limiting toxicity. Group 2 will continue to receive Tarceva 100mg/day po. All patients will continue to receive gemcitabine 1000mg/m2 iv on days 1, 8 and 15 of each 4 week cycle. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* histologically or cytologically confirmed pancreatic cancer with measurable or non-measurable metastatic disease;
* ECOG performance status of 0-1.

Exclusion Criteria:

* local, or locally advanced, pancreatic cancer;
* prior systemic treatment for metastatic pancreatic cancer;
* <=6 months since last adjuvant chemotherapy;
* other malignancies within last 5 years, except for adequately treated cancer in situ of the cervix, or basal or squamous cell skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 467 (Actual)
Dates: Start 2008-05; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (82):
- Argentina (4):
  - Buenos Aires
  - Rosario
  - San Juan Bautista
  - Santa Fe
- Australia (8):
  - Canberra, Australian Capital Territory
  - Liverpool, New South Wales
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Brisbane, Queensland
  - Adelaide, South Australia
  - Ballarat, Victoria
  - Frankston, Victoria
- Austria (2):
  - Salzburg
  - Vienna
- Belgium (5):
  - Antwerp
  - Brussels
  - Ghent
  - Leuven
  - Liège
- Brazil (5):
  - Salvador, Estado de Bahia
  - Belo Horizonte, Minas Gerais
  - Ijuí, Rio Grande do Sul
  - Santo André, São Paulo
  - São Paulo, São Paulo
- Canada (2):
  - Mississauga, Ontario
  - Toronto, Ontario
- Zagreb, Croatia
- Denmark (3):
  - Copenhagen
  - Herlev
  - Hillerød
- France (5):
  - Angers
  - Besançon
  - Brest
  - Paris
  - Saint-Priest-en-Jarez
- Germany (15):
  - Berlin
  - Bochum
  - Bonn
  - Esslingen am Neckar
  - Halle
  - Hamburg
  - Hamm
  - Kaiserslautern
  - Leipzig
  - Marburg
  - Mönchengladbach
  - München
  - Saarbrücken
  - Trier
  - Ulm
- Greece (2):
  - Heraklion
  - Thessaloniki
- Hong Kong, Hong Kong
- Israel (5):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Aviv
  - Ẕerifin
- Italy (7):
  - Chieti, Abruzzo
  - San Giovanni Rotondo, Apulia
  - Napoli, Campania
  - Pordenone, Friuli Venezia Giulia
  - Udine, Friuli Venezia Giulia
  - Orbassano, Piedmont
  - Florence, Tuscany
- Vilnius, Lithuania
- Distrito Federal, Mexico
- Poland (4):
  - Gliwice
  - Lublin
  - Poznan
  - Warsaw
- Romania (4):
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Sibiu
- Serbia (2):
  - Belgrade
  - Kamenitz
- Singapore, Singapore
- Madrid, Madrid, Spain
- Taipei, Taiwan
- United Kingdom (2):
  - London
  - Salisbury

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine (G) Plus (+) Erlotinib (E): Rash ≥ Grade 2: Participants began a 4 week run-in period where they received gemcitabine, 1000 milligrams per square meter (mg/m^2), intravenously (IV), on Days 1, 8, 15, 22 until development of a rash Grade ≥ 2. Participants also received erlotinib, 100 milligrams (mg), orally (PO) as a film-coated tablet, once daily until development of a rash Grade ≥ 2. Participants were not randomized to a treatment arm, but continued to receive the standard treatment of gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of consecutive 4 week cycles, and erlotinib, 100 mg, PO as a film-coated tablet, once daily until disease progression, unacceptable toxicity, or withdrawal for up to 46 months.
- G+E Standard Dose: Rash Grade Less Than (<) 2: Participants completed a 4 week run-in period where they received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, 15, 22. Participants also received erlotinib, 100 mg, PO as a film-coated tablet, once daily for 4 weeks. Participants without evidence of clinical progression and who had not developed rash Grade ≥ 2 or any other toxicity leading to dose adjustments or discontinuation were randomized to receive gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of consecutive 4 week cycles and erlotinib, 100 mg, PO as a film-coated tablet, once daily until disease progression or unacceptable toxicity, or withdrawal for up to 46 months.
- G+E Escalating Dose: Rash Grade < 2: Participants completed a 4 week run-in period where they received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, 15, 22. Participants also received erlotinib, 100 mg, PO as a film-coated tablet, once daily for 4 weeks. Participants without evidence of clinical progression and who had not developed rash Grade ≥ 2 or any other toxicity leading to dose adjustments or discontinuation were randomized to receive erlotinib, beginning at 150 milligrams per day (mg/day), PO as a film-coated tablet, once daily and increasing in increments of 50 mg every 2 weeks up to a maximum of 250 mg/day, until development of a Grade ≥ 2 rash, or occurrence of other, non-rash, dose-limiting toxicity; treatment was continued until disease progression, unacceptable toxicity, death or withdrawal for up to 46 months. Those participants also received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of consecutive 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for up to 46 months.
- G+E: No Rash Non-Eligibl: Participants began a 4 week run-in period where they received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, 15, 22 until the appearance of evidence of clinical progression or other toxicity leading to dose adjustments or discontinuation. Participants also received erlotinib, 100 mg, PO as a film-coated tablet, once daily until the appearance of evidence of clinical progression or other toxicity leading to dose adjustments or discontinuation. Participants were not randomized to a treatment arm, but continued to receive the standard treatment of gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of consecutive 4 week cycles, and erlotinib, 100 mg, PO as a film-coated tablet, once daily until disease progression, unacceptable toxicity, or withdrawal for up to 46 months.
- G+E: Early Drop Out: Participants began a 4 week run-in period where they received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, 15, 22 for up to 4 weeks. Participants also received erlotinib, 100 mg, PO as a film-coated tablet, once daily for up to 4 weeks.
Period: Overall Study
Arm/Group | Gemcitabine (G) Plus (+) Erlotinib (E): Rash ≥ Grade 2 | G+E Standard Dose: Rash Grade Less Than (<) 2 | G+E Escalating Dose: Rash Grade < 2 | G+E: No Rash Non-Eligibl | G+E: Early Drop Out
Started | 106 | 75 | 71 | 179 | 36
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 106 | 75 | 71 | 179 | 36
Not completed — Adverse Event | 8 | 4 | 7 | 17 | 13
Not completed — Death | 5 | 4 | 1 | 8 | 5
Not completed — Lack of Efficacy | 84 | 58 | 53 | 133 | 13
Not completed — Violation of Selection Criteria | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Refused treatment | 3 | 7 | 6 | 17 | 5
Not completed — Other | 5 | 2 | 3 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis population (SAP): all participants who received at least 1 dose of the trial medication and had at least 1 safety follow-up, whether withdrawn prematurely or not.
Groups:
- G+E: Rash ≥ Grade 2: Participants began a 4 week run-in period where they received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, 15, 22 until development of a rash Grade ≥ 2. Participants also received erlotinib, 100 mg, PO as a film-coated tablet, once daily until development of a rash Grade ≥ 2. Participants were not randomized to a treatment arm, but continued to receive the standard treatment of gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of consecutive 4 week cycles, and erlotinib, 100 mg, PO as a film-coated tablet, once daily until disease progression, unacceptable toxicity, or withdrawal for up to 46 months.
- G+E Standard Dose: Rash Grade < 2: Participants completed a 4 week run-in period where they received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, 15, 22. Participants also received erlotinib, 100 mg, PO as a film-coated tablet, once daily for 4 weeks. Participants without evidence of clinical progression and who had not developed rash Grade ≥ 2 or any other toxicity leading to dose adjustments or discontinuation were randomized to receive gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of consecutive 4 week cycles and erlotinib, 100 mg, PO as a film-coated tablet, once daily until disease progression or unacceptable toxicity, or withdrawal for up to 46 months.
- G+E Escalating Dose: Rash Grade < 2: Participants completed a 4 week run-in period where they received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, 15, 22. Participants also received erlotinib, 100 mg, PO as a film-coated tablet, once daily for 4 weeks. Participants without evidence of clinical progression and who had not developed rash Grade ≥ 2 or any other toxicity leading to dose adjustments or discontinuation were randomized to receive erlotinib, beginning at 150 mg/day, PO as a film-coated tablet, once daily and increasing in increments of 50 mg every 2 weeks up to a maximum of 250 mg/day, until development of a Grade 2 rash, or occurrence of other, non-rash, dose-limiting toxicity; treatment was continued until disease progression, unacceptable toxicity, death or withdrawal for up to 46 months. Those participants also received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of consecutive 4 week cycles until disease progression, unacceptable toxicity, or withdrawal for up to 46 months.
- G+E: No Rash Non-Eligible: Participants began a 4 week run-in period where they received gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, 15, 22 until the appearance of evidence of clinical progression or other toxicity leading to dose adjustments or discontinuation. Participants also received erlotinib, 100 mg, PO as a film-coated tablet, once daily until the appearance of evidence of clinical progression or other toxicity leading to dose adjustments or discontinuation. Participants were not randomized to a treatment arm, but continued to receive the standard treatment of gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of consecutive 4 week cycles, and erlotinib, 100 mg, PO as a film-coated tablet, once daily until disease progression, unacceptable toxicity, or withdrawal for up to 46 months.
- Total: Total of all reporting groups
Arm/Group | G+E: Rash ≥ Grade 2 | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2 | G+E: No Rash Non-Eligible | G+E: Early Drop Out | Total
Number analyzed (Participants) | 106 | 75 | 70 | 179 | 36 | 466
Age, Customized [Number; unit: participants]
  Less Than (<) 65 Years | 66 | 43 | 34 | 97 | 21 | 261
  ≥ 65 Years | 40 | 32 | 36 | 82 | 15 | 205
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 41 | 34 | 77 | 15 | 208
  Male | 65 | 34 | 36 | 102 | 21 | 258

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Died Assessed From Point of Randomization
Description: Overall survival (OS) assessed from the point of randomization was defined as the time from randomization to the date of death due to any cause. Participants still alive at the time of analysis were censored at the date they were last known to be alive.
Time Frame: Randomization [Day 1 of Cycle 2 (4-week cycles)] and weekly thereafter for up to 46 months.
Population: Full analysis set (FAS): all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 75 | 70
percentage of participants | 81.3 | 85.7

2. Primary Outcome: OS Assessed From Point of Randomization
Description: OS assessed from the point of randomization was defined as the median time, in months, from randomization to the date of death due to any cause. Participants still alive at the time of analysis were censored at the date they were last known to be alive. The 95 percent (%) confidence interval (CI) was determined using Kaplan-Meier methodology.
Time Frame: Randomization [Day 1 of Cycle 2 (4-week cycles)] and weekly thereafter for up to 46 months.
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 75 | 70
months | 8.4 [6.4 to 10.0] | 7.0 [5.8 to 8.3]
Statistical Analysis 1: Comparison: G+E Standard Dose: Rash Grade < 2 vs G+E Escalating Dose: Rash Grade < 2; Test type: Superiority or Other; p = 0.2026, Log Rank; Hazard Ratio (HR) = 1.26, 95% CI 2-sided [0.88 to 1.80]

3. Secondary Outcome: Percentage of Participants With Disease Progression or Death as Assessed From Point of Randomization
Description: Progression-free survival (PFS) as assessed from the point of randomization was defined as the time from randomization to the first occurrence of progressive disease (PD) according to the Response Evaluation Criteria in Solid Tumors (RECIST) or death due to any cause. For target lesions (TLs), PD was defined as at least a 20% increase in the sum of longest diameter (SLD) of TLs, taking as reference the smallest SLD recorded since the treatment started. For non-target lesions (NTLs), PD was defined as unequivocal progression of existing NTLs. Participants who had neither progressed nor died at time of analysis were censored at the date of last tumor assessment.
Time Frame: Randomization [Day 1 of Cycle 2 (4-week cycles)] and weekly thereafter for up to 46 months.
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 75 | 70
percentage of participants | 90.7 | 88.6

4. Secondary Outcome: PFS Assessed From Point of Randomization
Description: PFS assessed from the point of randomization was defined as the median time, in weeks, from randomization to disease progression or death due to any cause. Participants who had neither progressed nor died at time of analysis were censored at the date of last tumor assessment. The 95% CI was determined using Kaplan-Meier methodology.
Time Frame: Randomization [Day 1 of Cycle 2 (4-week cycles)] and weekly thereafter for up to 46 months.
Population: FAS
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 75 | 70
weeks | 19.4 [16.0 to 26.9] | 15.3 [11.3 to 19.1]
Statistical Analysis 1: Comparison: G+E Standard Dose: Rash Grade < 2 vs G+E Escalating Dose: Rash Grade < 2; Test type: Superiority or Other; p = 0.6298, Log Rank; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.77 to 1.54]

5. Secondary Outcome: Percentage of Participants With a Best Overall Response (BOR) of Confirmed Complete Response (CR) or Partial Response (PR) According to RECIST
Description: BOR was defined as a confirmed CR or PR for at least 4 weeks. CR was defined as the disappearance of all TLs. PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the baseline (BL) SLD. The 95% CI for one sample binomial was determined using Pearson-Clopper method.
Time Frame: BL, Weeks 8, 16, 24, 32, 40, every 12 weeks thereafter until disease progression for up to 46 months.
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 75 | 70
percentage of participants | 14.7 [7.6 to 24.7] | 8.6 [3.2 to 17.7]
Statistical Analysis 1: Comparison: G+E Standard Dose: Rash Grade < 2 vs G+E Escalating Dose: Rash Grade < 2; Test type: Superiority or Other; p = 0.2543, Chi-squared; Difference in Response Rates = -6.10, 95% CI 2-sided [-17.2 to 5.0] — Approximate 95% CI for the difference of two rates was determined using the Hauck-Anderson method
Statistical Analysis 2: Comparison: G+E Standard Dose: Rash Grade < 2 vs G+E Escalating Dose: Rash Grade < 2; Test type: Superiority or Other; Odds Ratio (OR) = 0.55, 95% CI 2-sided [0.19 to 1.56]

6. Secondary Outcome: Percentage of Participants With a CR, PR, Stable Disease (SD), or PD According to RECIST
Description: CR was defined as the disappearance of all TLs. PR was defined as at least a 30% decrease in the SLD of the TLs, taking as a reference the BL SLD SD was defined as neither sufficient decrease in SLD to qualify for PR nor sufficient increase in SLD to qualify for PD. PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since the treatment started. The 95% CI for one sample binomial was determined using the Pearson-Clopper method.
Time Frame: BL, Weeks 8, 16, 24, 32, 40, every 12 weeks thereafter until disease progression for up to 46 months.
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 75 | 70
percentage of participants
  CR | 0.0 [0.0 to 4.8] | 1.4 [0.0 to 7.7]
  PR | 14.7 [7.6 to 24.7] | 7.1 [2.4 to 15.9]
  SD | 58.7 [46.7 to 69.9] | 72.9 [60.9 to 82.8]
  PD | 25.3 [16.0 to 36.7] | 12.9 [6.1 to 23.0]
  Missing (no response assessment) | 1.3 [NA to NA] — 95% CI was not determined for missing responses. | 5.7 [NA to NA] — 95% CI was not determined for missing responses.

7. Secondary Outcome: Percentage of Participants With SD (Maintained for at Least 8 Weeks) or CR or PR (Maintained for at Least 4 Weeks) According to RECIST
Description: Disease control was defined as a participant with a response of CR or PR for at least 4 weeks at any time during treatment, or SD that was maintained for at least 8 weeks after the start of treatment. The 95% CI for one sample binomial was determined using the Pearson-Clopper method.
Time Frame: BL, Weeks 8, 16, 24, 32, 40, every 12 weeks thereafter until disease progression for up to 46 months.
Population: FAS
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 75 | 70
percentage of participants | 62.7 [50.7 to 73.6] | 47.1 [35.1 to 59.4]
Statistical Analysis 1: Comparison: G+E Standard Dose: Rash Grade < 2 vs G+E Escalating Dose: Rash Grade < 2; Test type: Superiority or Other; p = 0.0603, Chi-squared; Difference in Disease Control Rates = -15.52, 95% CI 2-sided [-32.4 to 1.3] — Approximate 95% CI for the difference of two rates was determined using the Hauck-Anderson method

8. Secondary Outcome: Percentage of Participants Who Died as Assessed From Start of 4-Week Run-In
Description: OS assessed from the start of the 4-week run in period was defined as the time from BL to the date of death due to any cause. Participants still alive at the time of analysis were censored at the date they were last known to be alive.
Time Frame: BL and weekly thereafter for up to 46 months.
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | G+E: Rash ≥ Grade 2 | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 106 | 75 | 70
percentage of participants | 84.9 | 81.3 | 85.7

9. Secondary Outcome: OS Assessed From Start of 4-Week Run-In
Description: OS assessed from the start of the 4-week run in period was defined as the median time, in months, from BL to the date of death, due to any cause. Participants who were still alive at the time of analysis were censored at the date they were last known to be alive. The 95% CI was determined using Kaplan-Meier methodology.
Time Frame: BL and weekly thereafter for up to 46 months.
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | G+E: Rash ≥ Grade 2 | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 106 | 75 | 70
months | 7.9 [7.1 to 8.8] | 9.3 [7.3 to 10.9] | 8.0 [6.8 to 9.2]
Statistical Analysis 1: Comparison: G+E: Rash ≥ Grade 2 vs G+E Standard Dose: Rash Grade < 2; Test type: Superiority or Other; p = 0.2678, Log Rank; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.60 to 1.15]
Statistical Analysis 2: Comparison: G+E: Rash ≥ Grade 2 vs G+E Escalating Dose: Rash Grade < 2; Test type: Superiority or Other; p = 0.8449, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.74 to 1.43]

10. Secondary Outcome: Percentage of Participants With Disease Progression or Death as Assessed From the Start of 4-Week Run-In
Description: PFS as assessed from the start of 4-week run-in was defined as the time from BL to the first occurrence of PD according to RECIST or death due to any cause. For TLs, PD was defined as at least a 20% increase in the SLD of TLs, taking as reference the smallest SLD recorded since the treatment started. For NTLs, PD was defined as unequivocal progression of existing NTLs. Participants who had neither progressed nor died at time of analysis were censored at the date of last tumor assessment.
Time Frame: BL, Weeks 8, 16, 24, 32, 40, every 12 weeks thereafter until disease progression or death for up to 46 months.
Population: FAS
Measure: Number; unit: percentage of participants
Arm/Group | G+E: Rash ≥ Grade 2 | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 106 | 75 | 70
percentage of participants | 90.6 | 90.7 | 88.6

11. Secondary Outcome: PFS Assessed From the Start of 4-Week Run-In
Description: PFS assessed from the start of 4-week run-in was defined as the median time, in weeks, from BL to disease progression or death due to any cause. Participants who had neither progressed nor died at time of analysis were censored at the date of last tumor assessment. The 95% CI was determined using Kaplan-Meier methodology.
Time Frame: BL, Weeks 8, 16, 24, 32, 40, every 12 weeks thereafter until disease progression or death for up to 46 months.
Population: FAS; only participants with an event of PD or death were included in the analysis.
Measure: Median (95% Confidence Interval); unit: weeks
Groups:
- G+E: Rash ≥ Grade 2: Participants began a 4 week run-in period where they received gemcitabine, 1000 milligrams per square meter (mg/m^2), intravenously (IV), on Days 1, 8, 15, 22 until development of a rash Grade ≥ 2. Participants also received erlotinib, 100 milligrams (mg), orally (PO) as a film-coated tablet, once daily until development of a rash Grade ≥ 2. Participants were not randomized to a treatment arm, but continued to receive the standard treatment of gemcitabine, 1000 mg/m^2, IV, on Days 1, 8, and 15 of consecutive 4 week cycles, and erlotinib, 100 mg, PO as a film-coated tablet, once daily until disease progression, unacceptable toxicity, or withdrawal for up to 46 months.
Arm/Group | G+E: Rash ≥ Grade 2 | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2
Number analyzed (Participants) | 96 | 68 | 62
weeks | 17.1 [16.0 to 22.7] | 23.4 [20.0 to 31.0] | 19.3 [15.3 to 23.1]
Statistical Analysis 1: Comparison: G+E: Rash ≥ Grade 2 vs G+E Standard Dose: Rash Grade < 2; Test type: Superiority or Other; p = 0.0217, Log Rank; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.51 to 0.95]
Statistical Analysis 2: Comparison: G+E: Rash ≥ Grade 2 vs G+E Escalating Dose: Rash Grade < 2; Test type: Superiority or Other; p = 0.1596, Log Rank; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.57 to 1.10]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected up to 28 days after discontinuation of study drug, drug-related serious AEs (SAEs) continued to be collected thereafter.
Description: All participants who received at least 1 dose of trial medication and had at least 1 safety follow-up were included in the safety analysis population.
Arm/Group | G+E: Rash ≥ Grade 2 | G+E Standard Dose: Rash Grade < 2 | G+E Escalating Dose: Rash Grade < 2 | G+E: No Rash Non-Eligible | G+E: Early Drop Out
Serious Adverse Events (participants affected / at risk) | 39/105 | 24/77 | 20/71 | 64/178 | 22/36
Other Adverse Events (participants affected / at risk) | 105/105 | 74/77 | 71/71 | 178/178 | 34/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | G+E: Rash ≥ Grade 2 (N=105) | G+E Standard Dose: Rash Grade < 2 (N=77) | G+E Escalating Dose: Rash Grade < 2 (N=71) | G+E: No Rash Non-Eligible (N=178) | G+E: Early Drop Out (N=36)
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 1 | 4 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 4 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1 | 1 | 5 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 5 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Jejunal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0
Face injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Paraganglion neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 2 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 2 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 2 | 1 | 6 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 4 | 0
Sepsis (Infections and infestations) | 2 | 0 | 0 | 3 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 2 | 0
Biliary sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Biliary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Febrile infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Superinfection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 2 | 6 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 3 | 2 | 3 | 9 | 2
General physical health deterioration (General disorders) | 2 | 1 | 1 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 1 | 1
Death (General disorders) | 0 | 0 | 0 | 0 | 1
Device occlusion (General disorders) | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Sudden death (General disorders) | 0 | 0 | 0 | 0 | 1
Ulcer haemorrhage (General disorders) | 0 | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 1 | 2 | 3 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 2 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 2 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 2 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 2
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Sensory loss (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 2 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 1 | 0 | 0
Axillary vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Embolism venous (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | G+E: Rash ≥ Grade 2 (N=105) | G+E Standard Dose: Rash Grade < 2 (N=77) | G+E Escalating Dose: Rash Grade < 2 (N=71) | G+E: No Rash Non-Eligible (N=178) | G+E: Early Drop Out (N=36)
Diarrhoea (Gastrointestinal disorders) | 49 | 33 | 35 | 71 | 9
Nausea (Gastrointestinal disorders) | 50 | 28 | 24 | 69 | 9
Vomiting (Gastrointestinal disorders) | 27 | 17 | 23 | 43 | 8
Abdominal pain (Gastrointestinal disorders) | 26 | 13 | 16 | 49 | 3
Constipation (Gastrointestinal disorders) | 23 | 11 | 15 | 35 | 4
Abdominal pain upper (Gastrointestinal disorders) | 10 | 6 | 5 | 20 | 3
Ascites (Gastrointestinal disorders) | 3 | 3 | 2 | 8 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 47 | 18 | 15 | 78 | 8
Anaemia (Blood and lymphatic system disorders) | 26 | 26 | 27 | 66 | 10
Neutropenia (Blood and lymphatic system disorders) | 40 | 20 | 17 | 75 | 3
Leukopenia (Blood and lymphatic system disorders) | 8 | 7 | 3 | 29 | 1
Rash (Skin and subcutaneous tissue disorders) | 105 | 60 | 64 | 123 | 19
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 7 | 10 | 23 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 4 | 13 | 16 | 1
Fatigue (General disorders) | 32 | 17 | 23 | 53 | 3
Pyrexia (General disorders) | 29 | 22 | 15 | 44 | 6
Asthenia (General disorders) | 10 | 10 | 12 | 29 | 6
Oedema peripheral (General disorders) | 15 | 13 | 6 | 29 | 1
Mucosal inflammation (General disorders) | 10 | 8 | 8 | 15 | 2
Decreased appetite (Metabolism and nutrition disorders) | 31 | 17 | 24 | 52 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 4 | 9 | 10 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 7 | 7 | 20 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 7 | 3 | 17 | 3
Weight decreased (Investigations) | 9 | 7 | 15 | 22 | 1
Alanine aminotransferase increased (Investigations) | 4 | 6 | 5 | 7 | 4
Insomnia (Psychiatric disorders) | 13 | 8 | 8 | 14 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 7 | 10 | 9 | 0
Headache (Nervous system disorders) | 2 | 8 | 4 | 6 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 2 | 5 | 12 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 10 | 5 | 7 | 8 | 2
Dyspepsia (Gastrointestinal disorders) | 10 | 3 | 3 | 9 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 1 | 5 | 12 | 0
Aspartate aminotransferase increased (Investigations) | 5 | 4 | 2 | 9 | 3
Gamma-glutamyltransferase increased (Investigations) | 3 | 5 | 5 | 7 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 4 | 3 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 11 | 0
Depression (Psychiatric disorders) | 5 | 4 | 2 | 12 | 1
Anxiety (Psychiatric disorders) | 3 | 4 | 1 | 5 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 1 | 6 | 3
Deep vein thrombosis (Vascular disorders) | 3 | 4 | 3 | 3 | 2
Hypertension (Vascular disorders) | 5 | 5 | 3 | 5 | 0
General physical health deterioration (General disorders) | 4 | 2 | 4 | 2 | 0
Influenza like illness (General disorders) | 7 | 2 | 2 | 5 | 0
Pain (General disorders) | 2 | 4 | 4 | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4 | 7 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 0 | 2
Dizziness (Nervous system disorders) | 5 | 2 | 5 | 12 | 1
Dysgeusia (Nervous system disorders) | 6 | 4 | 7 | 7 | 0
Urinary tract infection (Infections and infestations) | 8 | 2 | 1 | 13 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.